CLINICAL TRIAL: NCT04512209
Title: Characterization of Biophysical Stromal Properties in Human Cancer: Towards Personalized Computational Oncology
Acronym: DCE-MRI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EC/2019/1330 (BC-06058)
Record Dates: First submitted 2020-07-31; First posted 2020-08-13 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Carcinomatosis, Peritoneal; Pancreas Cancer; Ovarian Cancer; Colon Cancer
MeSH Terms: conditions — Peritoneal Neoplasms; Pancreatic Neoplasms; Ovarian Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DCE-MRI (Experimental)
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI — Patients will undergo an MR scan before undergoing cytoreductive surgery. If neoadjuvant chemotherapy is administered, an extra MR scan is planned before the start of the neoadjuvant chemotherapy.
  During surgery, tissue samples will be taken for interstitial fluid pressure (IFP) measurement, immunohistochemistry (IHC) and characterization of biophysical properties (viscoelastic properties and hydraulic conductivity).

SUMMARY:
Drug delivery in solid tumors, whether administered systemically or locoregionally, is hindered by an elevated interstitial fluid pressure (IFP). Stromal targeting therapies are in active development, aiming to enhance drug transport after systemic or locoregional delivery. To date, no clinical methods are available to quantify tumor biophysical properties (including IFP). The investigators aim to use a combination of dynamic contrast enhanced MRI and computational fluid modeling (CFD) to measure stromal IFP in patients with pancreatic cancer and in patients with ovarian or colonic peritoneal carcinomatosis (PC). Computational data will be correlated with therapy response, platinum drug penetration, and invasively measured biophysical parameters after intravenous (pancreas) or intraperitoneal (ovarian/colonic PC) administration of a platinum compound. This would be the first in depth clinical study addressing this important topic, and could pave the way to developing personalized computational based treatment approaches aimed at targeting the biophysical environment of the tumor stroma in order to enhance cancer drug delivery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-cystic adenocarcinoma the pancreas requiring neoadjuvant chemotherapy (any) because of borderline resectability
* Patients with stage IIIC or IVA ovarian cancer planned for debulking and HIPEC.
* Patients with stage IIIC or IVA colorectal cancer planned for debulking and HIPEC

Exclusion Criteria:

* Age <18 years
* Pregnancy, or suspected inadequate contraception during study period
* Clinically detectable ascites
* Intestinal or urinary tract obstruction
* Hepatic and/or extra-abdominal metastatic disease
* Impaired renal function (serum creatinine > 1.5mg/dl or calculated GFR (CKD-EPI) < 60mL/min/1.73 m²)
* Impaired liver function (serum total bilirubin > 1.5 mg/dl, except for known Gilbert's disease)
* Platelet count < 100.000/µl
* Hemoglobin < 9g/dl
* Neutrophil granulocytes < 1.500/ml
* Irresectable or metastatic disease
* Contra-indication for contrast enhanced MRI

  * Known allergy or intolerance to Gadolinium based contrast agents
  * Severe claustrophobia
  * Patients with metallic foreign bodies (pacemaker, neurostimulator, pedicle screw, cerebral aneurysm clips…) that may dislodge in a strong magnetic field
* Frail and medically unfit patients (Karnofsky index < 60% and WHO Performance score 3 or 4)
* Estimated life expectancy < 12 months
* In case of ovarian/colon cancer: no visible peritoneal metastasis on CT scan
* Acute or chronic pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2019-10-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Biophysical properties of the tumor tissue - measurement of Young modulus to assess viscoelasticity | up to 1 week after surgery
  A flat-ended cylindrical indentation tip, with 5 mm diameter, will be attached to a load cell to indent the sample. After the initial contact, the control algorithm will drive the tip to indent a given depth (30% of sample's height) into the test material at a constant velocity (1 mm/s). After reaching the prescribed depth, the position of the indentation tip will be fixed at this value for a given amount of time (300 s) in order to start the stress relaxation process. Units: Pa = kg m-1 s-2
Biophysical properties of the tumor tissue - measurement of hydraulic conductivity | up to 1 week after surgery
  The hydraulic conductivity of samples will be measured by detecting the amount of fluid exchange through the sample due to a hydrostatic pressure gradient in a closed system. The system includes two EasyMount Ussing diffusion chambers placed in a 2-channel EasyMount stand (Physiologic Instruments, Inc.; San Diego, CA), pressure reservoirs (syringes), and a bubble tracker device for measuring the liquid exchange.
  The nominal hydraulic conductivity (K') will be calculated by:
  K'=〖(d/D)〗^2 L/ρgh ∆x/∆t Where L and D are the tissue thickness and tissue area (interface), d is the glass tube diameter, ρ is the liquid density, h is the liquid column height, g is the gravity acceleration, x is bubble displacement and t is time.

SECONDARY OUTCOMES:
CFD modeling | up to 12 months after surgery
  Develop and validate a computational fluid dynamics (CFD) model to calculate interstitial fluid pressure based on dynamic contrast enhanced (DCE)-MRI data. This approach is based on Darcy's law (v=-K∇P) with v the velocity and ∇P the pressure gradient. The boundary condition at the outer edge of the tumor will be set to equal the convective outflow velocity values (v), as calculated during DCE-MRI. Hydraulic conductivity values (K) will be based on the tissue sample measurements. Other operational parameters such as the fluid properties (e.g. viscosity of interstitial fluid) will be based on literature values.
Measurement of Pt penetration | up to 24 months after surgery
  Quantitative laser ablation-ICP-MS will be used to analyze platinum penetration/distribution in peritoneal metastases that are left in situ during IP drug delivery but resected after completion of the procedure. The pixel intensities will be bilinearily interpolated and the Pt penetration depth set at 50% of the maximum intensity values.

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No